CLINICAL TRIAL: NCT05510999
Title: A Randomized, Double-blind, Placebo-controlled, Study to Investigate the Efficacy of Graminex® Flower Pollen Extracts in Healthy Women With Urinary Incontinence.
Brief Title: The Efficacy of Graminex® Flower Pollen Extracts in Healthy Women With Urinary Incontinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Graminex LLC (Other)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19GUHG
Record Dates: First submitted 2022-08-18; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Urinary Incontinence
Keywords: Safety and efficacy; Urinary incontinence; Urinary leakage
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Participants will be instructed to take one (1) capsule twice daily before breakfast and dinner with a glass of water for 24 weeks beginning on the Day 1, the day after their baseline visit. If a dose is missed participants are instructed to take the missed dose with the next scheduled dose. Participants will be advised not to exceed 3 capsules daily.
  Interventions: Other: Placebo
- Water soluble pollen extract fraction (Experimental): The experimental product contains 180mg (360mg/day) of water soluble pollen extract fraction. Participants will be instructed to take one (1) capsule twice daily before breakfast and dinner with a glass of water for 24 weeks beginning on the Day 1, the day after their baseline visit. If a dose is missed participants are instructed to take the missed dose with the next scheduled dose. Participants will be advised not to exceed 3 capsules daily.
  Interventions: Dietary Supplement: Water soluble pollen extract fraction
- Lipid soluble pollen extract fraction + water soluble pollen extract fraction (Experimental): The experimental product is a combination of 9 mg lipid soluble pollen extract fraction (18mg/day) and 180 mg water soluble pollen extract fraction (360mg/day). Participants will be instructed to take one (1) capsule twice daily before breakfast and dinner with a glass of water for 24 weeks beginning on the Day 1, the day after their baseline visit. If a dose is missed participants are instructed to take the missed dose with the next scheduled dose. Participants will be advised not to exceed 3 capsules daily.
  Interventions: Dietary Supplement: Lipid soluble pollen extract fraction + water soluble pollen extract fraction
- Lipid soluble pollen extract fraction (Experimental): The experimental product contains 9mg (18mg/day) of lipid soluble pollen extract fraction. Participants will be instructed to take one (1) capsule twice daily before breakfast and dinner with a glass of water for 24 weeks beginning on the Day 1, the day after their baseline visit. If a dose is missed participants are instructed to take the missed dose with the next scheduled dose. Participants will be advised not to exceed 3 capsules daily.
  Interventions: Dietary Supplement: Lipid soluble pollen extract fraction
- Water soluble pollen extract fraction + cranberry powder (Experimental): The experimental product is a combination of 42 mg water soluble pollen extract fraction (84 mg/day) and 125 mg cranberry powder (250 mg/day). Participants will be instructed to take one (1) capsule twice daily before breakfast and dinner with a glass of water for 24 weeks beginning on the Day 1, the day after their baseline visit. If a dose is missed participants are instructed to take the missed dose with the next scheduled dose. Participants will be advised not to exceed 3 capsules daily.
  Interventions: Dietary Supplement: Water soluble pollen extract fraction + cranberry powder

INTERVENTIONS:
Other: Placebo — One capsule of placebo will be taken twice daily for 24 weeks.
  Arms: Placebo
Dietary Supplement: Water soluble pollen extract fraction — Each capsule contains 180 mg of water soluble pollen extract fraction. One capsule will be taken twice daily (360 mg/day) for 24 weeks.
  Arms: Water soluble pollen extract fraction
Dietary Supplement: Lipid soluble pollen extract fraction + water soluble pollen extract fraction — Each capsule contains a combination of 9 mg of lipid soluble pollen extract fraction and 180 mg of water soluble pollen extract fraction. One capsule will be taken twice daily (18 mg/day and 360 mg/day, respectively) for 24 weeks.
  Arms: Lipid soluble pollen extract fraction + water soluble pollen extract fraction
Dietary Supplement: Lipid soluble pollen extract fraction — Each capsule contains 9 mg of lipid soluble pollen extract fraction. One capsule of will be taken twice daily (18 mg/day) for 24 weeks.
  Arms: Lipid soluble pollen extract fraction
Dietary Supplement: Water soluble pollen extract fraction + cranberry powder — Each capsule contains a combination of 42 mg of water soluble pollen extract and 125 mg of cranberry powder. One capsule will be taken twice daily (84 mg/day and 250 mg/day, respectively) for 24 weeks.
  Arms: Water soluble pollen extract fraction + cranberry powder

SUMMARY:
The primary objective of this study is to investigate the effect of Graminex® Flower Pollen Extracts in healthy women with urinary incontinence. The change in severity of urinary incontinence between baseline and 24 weeks will be assessed by an International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), and compared between the investigational product and placebo groups. Additionally, the safety and tolerability of Graminex® Flower Pollen Extracts, as compared to placebo, will be measured by the occurrence of and/or changes in treatment-emergent adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Females between the ages of 40-75 inclusive.
2. BMI 18.5 kg/m2 - 34.9 kg/m2 inclusive.
3. Involuntary loss of urine (incontinence) persisting for at least 1 month as determined by a score ≥ 5 on the ICIQ-SF questionnaire at the screening visit.
4. Female participant is not of child-bearing potential, defined as females who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation) or have been post-menopausal (natural or surgically) for at least 1 year prior to screening.

   Or,

   Females of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
5. Agree to keep lifestyle habits consistent (dietary habits and physical activity patterns) for the duration of the trial.
6. Willing to maintain current caffeine intake. Individuals with excessive habitual caffeine intake (>3 cups coffee or >4 cups caffeinated tea per day or >2 energy drinks) will be required to reduce consumption for 2 weeks prior to baseline.
7. Healthy as determined by laboratory results, medical history, and physical exam.
8. Has given voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the trial.
2. Allergy or sensitivity to test product ingredients.
3. Treatment (ie. pessary) or surgery (ie. sling, mesh) for urinary incontinence from a continence specialist (ie. urologist, urogynecologist, gynecologist) within the past 5 years.
4. Treatment for overactive or neurogenic bladder in previous 3 months (ie. neuromodulation, botox).
5. Initiation of pelvic floor therapy in the previous 3 months.
6. Current utilization of a catheter for urination.
7. Current urinary tract infection (UTI, confirmed by laboratory analysis), verbal confirmation of infection in previous 3 months or history of recurrent UTIs.
8. Women who are currently taking medications for urinary incontinence/overactive bladder (see Section 6.3.1).
9. Irregular menstrual periods within the previous 6 months (less than 21 or greater than 33 days between cycles).
10. Women who are within 1-year postpartum.
11. Genital malformation (i.e. Vaginal fistula) or vaginal and/or vulvar disorder (i.e. vulvovaginal atrophy).
12. Women on hormone replacement therapy (oral or topical), unless on a stable dose for ≥6 months.
13. Metal implants that may affect the DXA scan results will be assessed on case-by-case basis by the QI.
14. Current, chronic constipation reviewed on a case-by-case basis by the QI.
15. Current or history of diabetes.
16. Current or history of bladder tumour.
17. Current sexually transmitted infection (confirmed by laboratory analysis), or verbal confirmation of infection in previous 3 months.
18. Current or history of liver, kidney or heart disease.
19. Current or pre-existing unstable thyroid condition. Treatment on a stable dose of medication for over one year will be reviewed on a case-by-case basis by the QI .
20. Current or history of bleeding disorders.
21. Clinically significant abnormal laboratory results at screening.
22. Excessive consumption of alcohol equivalent to >2 alcoholic drinks/day (average).
23. Alcohol or drug abuse within the last 6 months.
24. Individuals who are cognitively impaired and/or who are unable to give informed consent.
25. Any autoimmune disease or immune-compromised (i.e. HIV positive, use of anti-rejection medication, rheumatoid arthritis, Hepatitis B/C positive).
26. Participation in other clinical research trials one month prior to or during enrollment will be assessed case-by-case by the QI.
27. Any other condition, that, in the opinion of the QI, may adversely affect the participant's ability to provide written informed consent and complete the study or its measures, or pose significant risk to the participant.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
The change in severity of urinary incontinence between baseline and 24 weeks. | baseline and 24 weeks
  The change in severity of urinary incontinence between baseline and 24 weeks as assessed by the ICIQ-SF will be compared between groups assigned to the Graminex® Flower Pollen Extracts and placebo.

SECONDARY OUTCOMES:
The change in severity of urinary incontinence between baseline and week 6, 12, and 18. | baseline, week 6, week 12, week 18
  The change in severity of urinary incontinence between baseline and week 6, 12, and 18 as assessed by the ICIQ-SF will be compared between groups assigned to the Graminex® Flower Pollen Extracts and placebo.
The change in frequency of urinary incontinence between baseline and week 6, 12, 18, and 24. | baseline, week 6, week 12, week 18, week 24
  The change in frequency of urinary incontinence between baseline and week 6, 12, 18, and 24 as assessed by void diary will be compared between groups assigned to the Graminex® Flower Pollen Extracts and placebo.
The change in daily urinary leakage volume between baseline and week 6, 12, 18, and 24. | baseline, week 6, week 12, week 18, week 24
  The change in daily urinary leakage volume between baseline and week 6, 12, 18, and 24 as assessed by 24-hour pad weight will be compared between groups assigned to the Graminex® Flower Pollen Extracts and placebo.
The change in stress-induced urinary leakage volume between baseline and week 24. | baseline, week 24
  The change in stress-induced urinary leakage volume between baseline and week 24 as assessed by pad weight following a provocative maneuvers challenge will be compared between groups assigned to the Graminex® Flower Pollen Extracts and placebo.
The change in frequency of nocturia between baseline and week 6, 12, 18, and 24. | baseline, week 6, week 12, week 18, week 24
  The change in frequency of nocturia between baseline and week 6, 12, 18, and 24 as assessed by void diary will be compared between groups assigned to the Graminex® Flower Pollen Extracts and placebo.
The change in frequency of daytime urination between baseline and week 6, 12, 18, and 24. | baseline, week 6, week 12, week 18, week 24
  The change in frequency of daytime urination between baseline and week 6, 12, 18, and 24 as assessed by void diary will be compared between groups assigned to the Graminex® Flower Pollen Extracts and placebo.
The change in bone density between baseline and week 24. | baseline, week 24
  The change in frequency of bone density between baseline and week 24 as assessed by DXA scan will be compared between groups assigned to the Graminex® Flower Pollen Extracts and placebo.
The change in incontinence-related quality of life between baseline and weeks 6, 12, 18, and 24. | baseline, week 6, week 12, week 18, week 24
  The change in incontinence-related quality of life between baseline and weeks 6, 12, 18, and 24 as assessed by I-QoL will be compared between groups assigned to the Graminex® Flower Pollen Extracts and placebo.
The change in degree of bother between baseline and weeks 6, 12, 18, and 24. | baseline, week 6, week 12, week 18, week 24
  The change in degree of bother between baseline and weeks 6, 12, 18, and 24 as assessed by OAB-q will be compared between groups assigned to the Graminex® Flower Pollen Extracts and placebo.
The change in sleep quality between baseline and weeks 6, 12, 18, and 24. | baseline, week 6, week 12, week 18, week 24
  The change in sleep quality between baseline and weeks 6, 12, 18, and 24 as assessed by Sleep Index will be compared between groups assigned to the Graminex® Flower Pollen Extracts and placebo.
The change in Lower Urinary Tract Symptom Score (LUTSS) between baseline and weeks 6, 12, 18, and 24. | baseline, week 6, week 12, week 18, week 24
  The change in Lower Urinary Tract Symptom Score (LUTSS) between baseline and weeks 6, 12, 18, and 24 as assessed by the LUTSS Questionnaire will be compared between groups assigned to the Graminex® Flower Pollen Extracts and placebo.
The incidence of pre-emergent and post-emergent adverse events during a 24-week supplementation period. | 24 weeks
Vital sign measurements (blood pressure; BP) during a 24-week supplementation period. | baseline, week 6, week 12, week 18, week 24
Vital sign measurements (heart rate; HR) during a 24-week supplementation period. | baseline, week 6, week 12, week 18, week 24
Aspartate aminotransferase (AST) measurement following a 24-week supplementation. | 24 weeks
  Clinical chemistry (including aspartate aminotransferase (AST)) will be measured in blood from study participants at 24 weeks.
Alanine aminotransferase (ALT) measurement following a 24-week supplementation. | 24 weeks
  Clinical chemistry (including alanine aminotransferase (ALT)) will be measured in blood from study participants at 24 weeks.
Bilirubin measurement following a 24-week supplementation. | 24 weeks
  Clinical chemistry (including bilirubin) will be measured in blood from study participants at 24 weeks.
Creatinine measurement following a 24-week supplementation. | 24 weeks
  Clinical chemistry (including creatinine) will be measured in blood from study participants at 24 weeks.
Measurement of electrolytes following a 24-week supplementation. | 24 weeks
  Clinical chemistry (including electrolytes (Na, K, Cl,)) will be measured in blood from study participants at 24 weeks.
Estimated glomerular filtration rate (eGFR) measurements following a 24-week supplementation. | 24 weeks
  Clinical chemistry (including estimated glomerular filtration rate (eGFR)) will be measured in blood from study participants at 24 weeks.
White blood cell measurements following a 24-week supplementation. | 24 weeks
  Hematology measurements (including white blood cell count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils) will be measured in blood from study participants at 24 weeks.
Red blood cell measurements following a 24-week supplementation. | 24 weeks
  Hematology measurements (including red blood cell count) will be measured in blood from study participants at 24 weeks.
Hemoglobin measurements following a 24-week supplementation. | 24 weeks
  Hematology measurements (including hemoglobin) will be measured in blood from study participants at 24 weeks.
Hematocrit measurements following a 24-week supplementation. | 24 weeks
  Hematology measurements (including hematocrit) will be measured in blood from study participants at 24 weeks.
Platelet count measurements following a 24-week supplementation. | 24 weeks
  Hematology measurements (including platelet count) will be measured in blood from study participants at 24 weeks.
Mean corpuscular hemoglobin following a 24-week supplementation. | 24 weeks
  Red blood cell indices (including mean corpuscular hemoglobin) will be measured in blood from study participants at 24 weeks.
Mean corpuscular hemoglobin concentration following a 24-week supplementation. | 24 weeks
  Red blood cell indices (including mean corpuscular hemoglobin concentration) will be measured in blood from study participants at 24 weeks.
Mean corpuscular volume following a 24-week supplementation. | 24 weeks
  Red blood cell indices (including mean corpuscular volume) will be measured in blood from study participants at 24 weeks.
Red cell distribution width following a 24-week supplementation. | 24 weeks
  Red blood cell indices (including red cell distribution width) will be measured in blood from study participants at 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No